CLINICAL TRIAL: NCT01843608
Title: Effect of Combined Training Post-treatment Intervention in Lean Body Mass Recovery in Breast Cancer Survival. A Randomised Controlled Trial.
Brief Title: Effect of Combined Exercise Post-treatment Intervention in Lean Mass Recovery in Breast Cancer Survival.
Acronym: WIM1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Soraya Casla Barrio, PhD Student, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSMSCCMYEJ1
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Sarcopenic Obesity in Breast Cancer Survival; Muscle Strength Quantitative Trait Locus 1; Cardiopulmonary Capacity; Quality of Life; Fatigue; Depression
Keywords: Physical treatment; Exercise prescription to breast cancer survival; Side cancer effect treatment
MeSH Terms: conditions — Fatigue; Depression | interventions — Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients in this group will be asked to maintain the same activity level until the baseline assessments.
  They cannot change physical activity and nutritional habits.
- Physical Intervention Group (Experimental): They have to perform two days per week of guide and planned exercise during three months. All classes are composed by different parts: aerobic exercise, to improve cardiovascular capacity, strength, to work muscle mass and flexibility to increase joint movements.
  They have to present an attendance above or equal to 80%.
  Interventions: Other: Physical Intervention

INTERVENTIONS:
Other: Physical Intervention — The exercise program will be designed and conducted by qualified in Physical Activity and Sport Sciences. The exercise program will consist in a combined two days per week of supervised training program and one day per week of briskly walking by themselves, following a document, designed by the specialist trainer, which will be given at the beginning of the program. The intervention will have a duration of 12 consecutive weeks. The intensity will be increasing progressively from 65% to 85% of heart rate. The intensity will be controlled by heart rate monitor trademark POLAR FT7 in aerobic exercise and with the number of repetitions (from 8 to 15) and sets (from 2 to 3) in strength exercises. Prescription intensity will be done using Karvonen equation, recommended method to work with risk population.
  Other Names: Women In Motion
  Arms: Physical Intervention Group

SUMMARY:
Breast cancer survival it is affected by the side effects related to the illness, the treatments or even the behavioral factors (e.g. inadequate diet, sedentary behavior) that create in this women an important quantity of psychological and physical disorders. Prior systematic reviews and meta-analyses have demonstrate that supervised aerobic training is a safe, feasible, and effective adjunct therapy to improve a broad range of physiological and psychological outcomes in women with early breast cancer. However the vast majority of studies to date have focused on the efficacy of exercise to improve symptom control outcomes in breast cancer patients either during or following the completion of adjuvant therapy.

Most relevant consequences are found in women that have to undergo surgery as 16% to 43% of women with breast cancer suffer functional limitation in the shoulder, inflammation, pain or strength and flexibility reduction in upper body limbs one year after surgery with a high prevalence which is rising.

Weight gain is associated with decreased quality of life and increased risk for several comorbid conditions, such as cardiovascular disease and diabetes. The most of the cardiopulmonary problems are induced by chemotherapy or radiotherapy, because of the treatments effect in the heart and its consequences in cardiorespiratory fitness of these women.

These side effects become in important limitations to allow women return their normal life style. These limitations have a severe effect in decreasing of physical activity practice, which have visible consequences in increasing general fatigue and calcium deficiency in bones due to the age and some adjuvant treatments.

Previous studies found that patients with breast cancer who gained modest amounts of weight were significantly more likely to experience disease recurrence and die from breast cancer and other causes that those who were weight stable. In addition, two thirds of the studies that have assessed body composition change in relation to weight gain in this patient population observe no net gain in muscle mass or loss in muscle mass as body weight and adipose tissue increase. These changes are defined as sarcopenic obesity. This kind of obesity is characterized by weight gain in the presence of lean tissue loss or absence of lean tissue gain. In addition fat tissue gain is related with other health disorders such as diabetes, functional limitations and poor survival levels. Treatment for this unique pattern of weight gain is an exercise intervention, especially strength training.

Psychological effects have to be took account as cancer produce important aftermath. Large scientific evidence shows the psycho-emotional alterations in women diagnosed with breast cancer at some point in their life.

World Health Organization (WHO) defines quality of life as "individuals perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. It is a broad ranging concept affected in a complex way by the person's physical health, psychological state, level of independence, social relationships, personal beliefs and their relationship to salient features of their environment." Following this definition numbered of researches have been developed, presenting interest in both physiological and psychological changes and improvements, as show different studies.

HYPOTHESIS The primary hypothesis of this study is that group exercise intervention, combining aerobic and strength training, will reduce lean mass and body fat tissue in breast cancer post treatment survival.

Secondary hypothesis of this clinical trial are follows:

1. Combined exercise intervention will increase maximal strength level of chest press and leg press.
2. Combined exercise intervention will increase maximal cardiopulmonary capacity, assessed by Peak Oxygen Consumption(VO2peak), which has been confirmed as an important value in survivals. In addition, ACSM propose this value as the Gold Standard to assess fitness level.
3. Combined exercise intervention will increase global Isometric Strength Index, assessed by Grip Strength Dynamometer.
4. Combined exercise intervention will improve range motion in upper-limbs.
5. Patients Reported Outcomes (PROs), such as quality of life (QoL), Health perception and depression.

DETAILED DESCRIPTION:
This study will be a 3-month, two arms, randomized controlled exercise intervention trial, will be developed. After baseline measurements, participants will be randomized into the treatment and control groups by using a blocked randomization procedure.

This study will be developed through a collaboration between Technical University of Madrid (UPM) and Cancer Patients Spanish Group (GEPAC). This project will be carried out at the facilities of the Physical Activity and Sport Science (FCCAFD-INEF) and it was approved by the Ethical Committee of the UPM.

Women will be recruited from hospitals through posters and oncologist information and the diffusion of the project that GEPAC will do between their members. Women who present interest to be contacted will be phoned or mailed a study flyer and will be asked to fill in an initial questionnaire The intervention will be performed in a social framework. It will try to provide different skills to women, in order to improve self-trust and self-knowledge. Other important goal will be to give to women a space where they shared all their experiences and help women were going through the same situation.

The exercise program will be designed and conducted by qualified in Physical Activity and Sport Sciences. The exercise program will consist in a combined two days per week of supervised training program and one day per week of briskly walking by themselves, following a document, designed by the specialist trainer, which will be given at the beginning of the program. The intervention will have a duration of 12 consecutive weeks. The intensity will be increasing progressively from 65% to 85% of heart rate. The intensity will be controlled by heart rate monitor trademark POLAR FT7. Prescription intensity will be done using Karvonen equation, recommended method to work with risk population.

Every supervised session will have the same structure and will have a duration of 60 minutes. American College Sport Medicine (ACSM) Guidelines for Cancer Patients will be followed for the session design. Participants will be divided in groups of 15 per class to provide more individual attendance.

The first 10 minutes will be the warm up which will include joint mobilizations, different kinds of movements, briskly walking and running.

Next part will consist in aerobic exercise where the principal goal will be practice activities what will increase cardiopulmonary fitness and the functional capacity of the participants. Practiced activities will be "impact activities" which are the activities that weight is supported by the legs. They activate the bone regeneration and prevent osteoporosis. Interval training will be performed in this part, with 30 seconds of high intensity and 3 minutes of active recovery. Then, strength exercises with elastic band and activities where the women support the own weight will be developed to improve general strength and increase lean mass. The intensity will be quantified with the number of repetitions (from 8 to 15) and sets (from 2 to 3).

The last part will be stretching exercises dedicated to improve the joint mobility and the muscle flexibility of upper body limbs and the general muscles relax after training.

Women will be contacted 3 months after the project to know the real effect in adherence of the participant and in the global strength.

All adverse events that could occur during the intervention time will be register for the project coordinator contacting by phone with the patients.

These outcomes were assessed baseline and they were repeated after 12 weeks again.

Lean body mass and fat body mass Percentage of fat mass and percentage of muscle mas will be assessed by bio impedance, using TANITA BC-601F machine.

Demographics and clinical data Age, marital status, profession, quantity of physical activity before and after the disease, subtype of tumor, type of resection and type of endocrine medication will be recorded at baseline measurements.

Anthropometric assessments Weight, high, hip and waist circumferences and waist-hips ratio. Arm volumetries will be done to check that arm swelling did not increase.

Strength It will be assessed using two types of assessments. First type will be grip strength in hands, legs and back. Global strength will be assessed by Strength Index, which will be obtained adding all grip strength values and dividing de result by the participant weight. Grip Strength dynamomyter T.K.K.5401 to arms strength and T.K.K.5402 to legs and back strength will be used. Other studies will have used this method in order to obtain strength levels in breast cancer women demonstrating that is a feasible and safe method in this population. Second type of strength test will be 8 RM protocol to predict 1 Repetition Maximum (RM), following National Strength and Conditioning Association guidelines (NCSA 2008) and Mayhew formulae will be used to predict 1 RM. Test will be developed in PANATA machines.

Cardiovascular Capacity. It will be assessed by a submaximal cardiopulmonary exercise test following Prior to the start, women will have to complete the PAR-Q test to determine whether they are able to perform a graded exercise test.

Cardio-respiratory exercise responses will be assessed in each participant using a graded exercise test (GXT) on a treadmill. The test will be a modification of the Bruce GXT which was designed for use in clinical and older populations since the submaximal portion of the test can be done with walking and because it begins at a reduced intensity.

The ACSM guidelines to performance Cardio Pulmonary Exercise Test (CPET) will be followed to develop or to stop it, if it will be necessary.

Patient Report Outcomes

Quality of Life It is a very important outcome with a large definition related different concepts such as physical and psychological health, individual independence and social relationships. It was assessed by FACT-B questionnaire suggested in a review to be used in this population. The questionnaire presents 38 items and patients have to choose between 5 options (0 totally disagree and 4 totally agree) to describe their grade of accordance with the specific item

Depression Grade of depression was assessed by Center of Epidemiology Studies - Depression (CES.D). It was used in previous studies in order to determine the same outcome in breast cancer population. This test is a Likert scale, which presents 20 items. Patient has to identify how many times felt in that way during the previous week (from 0 never to 3 always). A score equal to 16 will be regarded as a mild depressive disorder

Health Survey Short Form -36 of Health Survey (SF-36) test will be used to assess Health Survey. Health status scores are abstractions, which obtain meaning through knowledge of how the scores are related to other variables and have been already used in cancer patients population. It presents 36 items and they are divided in 7 dimensions that will be interpreted together and separately.

Physical Activity Adherence and physical activity that women practice out of the program was collected by the validate questionnaire Godin Leisure-Time Test which registers times per week and intensity of the activities that women usually do in a typical week.

All statistical analyses will be done using SPSS Statistics 20.0 program. Confidential interval will be of 95% and the significance value will be 0.05 to determine the significance of the results.

Baseline characteristics of participants across the intervention and control groups were compared using Student t-test for continuous outcomes.

Between women comparisons of those randomized to treatment versus control for changes in FACT-B, FACT-F, SF-36 and CES-D, scores across months 0-3 will be made using Student t-test, after determining that adjustment for potential confounders do not alter the results.

Confounders examined included postmenopausal status, BMI status, baseline levels of sport and leisure-time physical activity.

Pearson correlation coefficients were used to evaluate associations between changes in body composition and strength and cardio-pulmonary status and changes in PROs scores. All probability values will be tested with the 2-tailed test.

Follow up 4 months after intervention will be compared with baseline and post intervention measures using ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosed confirmed stage I-IIIA.
* Randomized disposition.
* Minimum of forty-five days and maximum of thirty-six months after finishing treatments (chemotherapy and radiotherapy).
* 0-1 in Eastern Cooperative Oncology Group (ECOG) scale (present the ability to walk briskly)
* Oncologist approval.
* Informed Consent signed.
* Community of Madrid inhabitant.

Exclusion Criteria:

* Metastasis presence
* Serious medical risk such as unstable cardiac condition or severe pulmonary disease and anticoagulants treatments.
* Oncology or primary care approval who verified the medical risk exclusion criteria.
* ECOG > 1
* Pregnant

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Lean mass percentage | 3 months
  Lean body mass percentage in each participant before and after intervention in intervention group and three months after in control group, assessed by bioimpedance.
Maximal Strength | 3 months
  Maximal strength in upper limbs and in legs assessed by 8 RM protocol. Maxima resistance strength.

SECONDARY OUTCOMES:
Fat body mass | 3 months
  Percentage of body mass assessed by bio-impedance
Cardiovascular capacity | 3 months
  Submaximal cardiovascular capacity assessed by modified bruce protocol to 85% of maximal hearth rate.
Quality of Life | 3 moths
  Quality of Life level assessed by FACT-B Questionnaire. Each dimension will be analyzed separately.
Fatigue | 3 months
  Facit.org specific questionnaire will be used.
Health Perception | 3 months
  SF-36 questionnaire will be used.
Depression | 3 months
  CES-D questionnaire will be used and 16 will be the limit to define a depressive attitude.
Leisure-time exercise | 3 months
  It is the quantity of exercise that post treatment women do in them leisure-time and it is assessed by Godin Leisure-Time Exercise Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Sampedro, Professor, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Physical Activity and Sport Science Faculty, Madrid, Madrid, Spain

REFERENCES:
- [Background] Lacey JV Jr, Devesa SS, Brinton LA. Recent trends in breast cancer incidence and mortality. Environ Mol Mutagen. 2002;39(2-3):82-8. doi: 10.1002/em.10062. PMID 11921173
- [Background] Lopez-Abente G, Pollan M, Aragones N, Perez Gomez B, Hernandez Barrera V, Lope V, Suarez B. [State of cancer in Spain: incidence]. An Sist Sanit Navar. 2004 May-Aug;27(2):165-73. doi: 10.4321/s1137-66272004000300001. Spanish. PMID 15381948
- [Background] Chirlaque MD, Salmeron D, Ardanaz E, Galceran J, Martinez R, Marcos-Gragera R, Sanchez MJ, Mateos A, Torrella A, Capocaccia R, Navarro C. Cancer survival in Spain: estimate for nine major cancers. Ann Oncol. 2010 May;21 Suppl 3:iii21-29. doi: 10.1093/annonc/mdq082. PMID 20427356
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Lakoski SG, Eves ND, Douglas PS, Jones LW. Exercise rehabilitation in patients with cancer. Nat Rev Clin Oncol. 2012 Mar 6;9(5):288-96. doi: 10.1038/nrclinonc.2012.27. PMID 22392097
- [Background] Sagen A, Karesen R, Risberg MA. Physical activity for the affected limb and arm lymphedema after breast cancer surgery. A prospective, randomized controlled trial with two years follow-up. Acta Oncol. 2009;48(8):1102-10. doi: 10.3109/02841860903061683. PMID 19863217
- [Background] Chlebowski RT, Aiello E, McTiernan A. Weight loss in breast cancer patient management. J Clin Oncol. 2002 Feb 15;20(4):1128-43. doi: 10.1200/JCO.2002.20.4.1128. PMID 11844838
- [Background] Roca-Alonso L, Pellegrino L, Castellano L, Stebbing J. Breast cancer treatment and adverse cardiac events: what are the molecular mechanisms? Cardiology. 2012;122(4):253-9. doi: 10.1159/000339858. Epub 2012 Aug 17. PMID 22907032
- [Background] Jones LW, Courneya KS, Mackey JR, Muss HB, Pituskin EN, Scott JM, Hornsby WE, Coan AD, Herndon JE 2nd, Douglas PS, Haykowsky M. Cardiopulmonary function and age-related decline across the breast cancer survivorship continuum. J Clin Oncol. 2012 Jul 10;30(20):2530-7. doi: 10.1200/JCO.2011.39.9014. Epub 2012 May 21. PMID 22614980
- [Background] Irwin ML, Crumley D, McTiernan A, Bernstein L, Baumgartner R, Gilliland FD, Kriska A, Ballard-Barbash R. Physical activity levels before and after a diagnosis of breast carcinoma: the Health, Eating, Activity, and Lifestyle (HEAL) study. Cancer. 2003 Apr 1;97(7):1746-57. doi: 10.1002/cncr.11227. PMID 12655532
- [Background] Riggs BL, Khosla S, Melton LJ 3rd. A unitary model for involutional osteoporosis: estrogen deficiency causes both type I and type II osteoporosis in postmenopausal women and contributes to bone loss in aging men. J Bone Miner Res. 1998 May;13(5):763-73. doi: 10.1359/jbmr.1998.13.5.763. PMID 9610739
- [Background] Winer EP, Hudis C, Burstein HJ, Wolff AC, Pritchard KI, Ingle JN, Chlebowski RT, Gelber R, Edge SB, Gralow J, Cobleigh MA, Mamounas EP, Goldstein LJ, Whelan TJ, Powles TJ, Bryant J, Perkins C, Perotti J, Braun S, Langer AS, Browman GP, Somerfield MR. American Society of Clinical Oncology technology assessment on the use of aromatase inhibitors as adjuvant therapy for postmenopausal women with hormone receptor-positive breast cancer: status report 2004. J Clin Oncol. 2005 Jan 20;23(3):619-29. doi: 10.1200/JCO.2005.09.121. Epub 2004 Nov 15. PMID 15545664
- [Background] Kroenke CH, Chen WY, Rosner B, Holmes MD. Weight, weight gain, and survival after breast cancer diagnosis. J Clin Oncol. 2005 Mar 1;23(7):1370-8. doi: 10.1200/JCO.2005.01.079. Epub 2005 Jan 31. PMID 15684320
- [Background] Aslani A, Smith RC, Allen BJ, Pavlakis N, Levi JA. Changes in body composition during breast cancer chemotherapy with the CMF-regimen. Breast Cancer Res Treat. 1999 Oct;57(3):285-90. doi: 10.1023/a:1006220510597. PMID 10617305
- [Background] Ingram C, Brown JK. Patterns of weight and body composition change in premenopausal women with early stage breast cancer: has weight gain been overestimated? Cancer Nurs. 2004 Nov-Dec;27(6):483-90. doi: 10.1097/00002820-200411000-00008. PMID 15632788
- [Background] Cheney CL, Mahloch J, Freeny P. Computerized tomography assessment of women with weight changes associated with adjuvant treatment for breast cancer. Am J Clin Nutr. 1997 Jul;66(1):141-6. doi: 10.1093/ajcn/66.1.141. PMID 9209182
- [Background] Demark-Wahnefried W, Peterson BL, Winer EP, Marks L, Aziz N, Marcom PK, Blackwell K, Rimer BK. Changes in weight, body composition, and factors influencing energy balance among premenopausal breast cancer patients receiving adjuvant chemotherapy. J Clin Oncol. 2001 May 1;19(9):2381-9. doi: 10.1200/JCO.2001.19.9.2381. PMID 11331316
- [Background] Demark-Wahnefried W, Hars V, Conaway MR, Havlin K, Rimer BK, McElveen G, Winer EP. Reduced rates of metabolism and decreased physical activity in breast cancer patients receiving adjuvant chemotherapy. Am J Clin Nutr. 1997 May;65(5):1495-501. doi: 10.1093/ajcn/65.5.1495. PMID 9129482
- [Background] Ligibel JA, Campbell N, Partridge A, Chen WY, Salinardi T, Chen H, Adloff K, Keshaviah A, Winer EP. Impact of a mixed strength and endurance exercise intervention on insulin levels in breast cancer survivors. J Clin Oncol. 2008 Feb 20;26(6):907-12. doi: 10.1200/JCO.2007.12.7357. PMID 18281663
- [Background] Heber D, Ingles S, Ashley JM, Maxwell MH, Lyons RF, Elashoff RM. Clinical detection of sarcopenic obesity by bioelectrical impedance analysis. Am J Clin Nutr. 1996 Sep;64(3 Suppl):472S-477S. doi: 10.1093/ajcn/64.3.472S. PMID 8780366
- [Background] Irwin ML. Physical activity interventions for cancer survivors. Br J Sports Med. 2009 Jan;43(1):32-8. doi: 10.1136/bjsm.2008.053843. Epub 2008 Oct 23. PMID 18948351
- [Background] McNeely ML, Campbell KL, Rowe BH, Klassen TP, Mackey JR, Courneya KS. Effects of exercise on breast cancer patients and survivors: a systematic review and meta-analysis. CMAJ. 2006 Jul 4;175(1):34-41. doi: 10.1503/cmaj.051073. PMID 16818906
- [Background] Segal R, Evans W, Johnson D, Smith J, Colletta S, Gayton J, Woodard S, Wells G, Reid R. Structured exercise improves physical functioning in women with stages I and II breast cancer: results of a randomized controlled trial. J Clin Oncol. 2001 Feb 1;19(3):657-65. doi: 10.1200/JCO.2001.19.3.657. PMID 11157015
- [Background] Demark-Wahnefried W, Case LD, Blackwell K, Marcom PK, Kraus W, Aziz N, Snyder DC, Giguere JK, Shaw E. Results of a diet/exercise feasibility trial to prevent adverse body composition change in breast cancer patients on adjuvant chemotherapy. Clin Breast Cancer. 2008 Feb;8(1):70-9. doi: 10.3816/CBC.2008.n.005. PMID 18501061
- [Background] Jones LW, Peppercom J, Scott JM, Battaglini C. Exercise therapy in the management of solid tumors. Curr Treat Options Oncol. 2010 Jun;11(1-2):45-58. doi: 10.1007/s11864-010-0121-5. PMID 20645033